CLINICAL TRIAL: NCT06250816
Title: The Effects of Wearing Operation Gown With Cartoon Characters on Reducing Preoperative Anxiety in Children: Randomized Controlled Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Selcan Akesen, MD, Uludag University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2023-28/21
Record Dates: First submitted 2023-12-20; First posted 2024-02-09 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Anxiety, Preoperative
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Children wearing the hospital gown with cartoon characters (Experimental): The experimental group will have a preoperative visit, the investigator will meet the patient and assess the child's anxiety level using the modified Yale Preoperative Anxiety Scale (m-YPAS). Afterwards, the patient will be asked to choose one of the hospital gowns they want to wear and put it on with parental assistance.
  Interventions: Other: The hospital gown with cartoon characters
- Children with standard hospital gown (No Intervention): The control group will have a preoperative visit, the investigator will meet the patient and assess the child's anxiety level using m-YPAS. The patient will be asked to wear the hospital gown used in the hospital in routine practice with parental assistance.

INTERVENTIONS:
Other: The hospital gown with cartoon characters — The patient will be asked to choose one of the hospital gowns with cartoon characters they want to wear and put it on with parental assistance.
  Arms: Children wearing the hospital gown with cartoon characters

SUMMARY:
The operating room environment can be frightening for pediatric patients. Many techniques have been used to make the operating room environment less intimidating, including allowing parents to accompany part of this procedure, play therapy and various distraction strategies during the entrance to the operating room. In a survey study, it was reported that parents were expected to create hospital conditions with a more child-friendly atmosphere. In this context, it is thought that creating a warmer environment for children, including the clothes worn in the operating room, may reduce the anxiety level of children. In this study, investigators' aim was to investigate the effect of wearing an hospital gown with cartoon characters on the reduction of preoperative anxiety in children scheduled for Orthopedic surgery by in the operating room.

DETAILED DESCRIPTION:
Pediatric patients aged between 4-12 years, who are planned to be operated by the Orthopedic Surgery Clinic in Bursa Uludag University Faculty of Medicine Hospital Surgical Theatre, will be randomized preoperatively by closed envelope method. One group will have a preoperative visit, the investigator will meet the patient and assess the child's anxiety level using the modified Yale Preoperative Anxiety Scale (m-YPAS). Afterwards, the patient will be asked to choose one of the hospital gowns they want to wear and put it on with parental assistance. The other group also will have a preoperative visit, the investigator will meet the patient and assess the child's anxiety level using m-YPAS. The patient will be asked to wear the hospital gown used in the hospital in routine practice with parental assistance. Then the patients will be taken to the operating room as in the routine procedure. Before induction of anesthesia in the operating room, another investigator will re-evaluate the child's anxiety level using the m-YPAS scale. Vital signs, analgesic use and duration of surgery will be recorded during the operation. Afterwards, the satisfaction level of the parents will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are planned to have elective orthopedic surgery
* Patients whose American Society of Anesthesiologists (ASA) physical status classification are between 1-3
* Patients who have approved the informed consent form

Exclusion Criteria:

* Motor and/or mentally retarded patients
* Patients with hearing-speech impairment
* Patients whose ASA physical status classification IV-V
* Patients who do not accept informed consent and/or refused to participate in the study

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
modified Yale Preoperative Anxiety Scale | 1 day
  investigators evaluate children using the verified Turkish version of modified Yale Preoperative Anxiety Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Selcan Akesen, MD, Principal Investigator — Uludağ Üniversitesi; Leman Gökçenur Aydın, MD, Study Director — Uludağ Üniversitesi
Locations (1):
- Uludağ Üniversitesi, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No